CLINICAL TRIAL: NCT00449605
Title: A Randomized, Double-Blind, Parallel-Group, Multicenter, Multinational Study to Assess Glycemic Control With Rimonabant in Comparison With Glimepiride Over 1 Year in Overweight/Obese Type2 Diabetic Patients Not Adequately Controlled With Metformin
Brief Title: A Glycemic Control Evaluation of Glimepiride Versus Rimonabant on Top of Metformin in Type 2 Diabetes
Acronym: ALLEGRO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC10007; 2006-005385-39 (EudraCT Number)
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Rimonabant; glimepiride; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rimonabant (Experimental): Rimonabant 20 mg once daily on top of metformin
  Interventions: Drug: Rimonabant; Drug: Metformin
- Glimepiride (Active Comparator): Glimepiride from 1 mg up to 6 mg once daily on top of metformin
  Interventions: Drug: Glimepiride; Drug: Metformin

INTERVENTIONS:
Drug: Rimonabant — Tablet, oral administration
  Other Names: SR141716; Acomplia
  Arms: Rimonabant
Drug: Glimepiride — Tablet, oral administration
  Other Names: HOE490; Amaryl
  Arms: Glimepiride
Drug: Metformin — Metformin continued at stable dose as background therapy

SUMMARY:
The primary objective is to demonstrate, after 52 weeks of treatment, the non-inferiority of rimonabant 20 mg once daily (od) versus glimepiride od in reducing glycosylated haemoglobin (HbA1c) in overweight/obese patients with type 2 diabetes not adequately controlled with metformin at a stable dose (≥ 1500 mg/day) for at least 3 months.

The main secondary objectives are to assess the effect of rimonabant in comparison with glimepiride on body weight and HDL-Cholesterol and the long-term safety and tolerability of rimonabant in comparison with glimepiride.

DETAILED DESCRIPTION:
The total duration per patient will be approximately 65 weeks including a 52-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with legal age
* Body Mass Index >27kg/m2
* Type 2 diabetes as defined by World Health Organization (WHO) criteria, treated with metformin for at least 6 months and with a stable dose of metformin >=1500 mg/day for at least three months
* HbA1c >=7% and <=9% at screening visit

Exclusion Criteria:

* Weight loss > 5 kg within three months prior to screening
* Presence of any clinically significant endocrine disease according to the Investigator
* Presence of type 1 diabetes
* Presence or history of cancer within the past 5 years with the exception of adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer
* Previous participation in a clinical study with rimonabant
* Absence of effective medical contraceptive method for females of childbearing potential
* Within 3 months prior to screening visit: use of oral antidiabetic drugs (other than metformin) and/or insulin, of anti-obesity drugs or other drugs for weight reduction
* Within 2 months prior to screening visit: administration of systemic long-acting corticosteroids or prolonged use (more than one week) of other systemic corticosteroids, change in lipid lowering treatment
* Presence of any severe medical or psychological condition or chronic conditions/infections that in the opinion of the Investigator would compromise the patient's safety or successful participation in the study, including uncontrolled serious psychiatric illness

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycemic measure HbA1c | 52 weeks (1 year)

SECONDARY OUTCOMES:
Absolute change from baseline in body weight | 52 weeks
Relative change from baseline in HDL-C | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (15):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Chile (2):
  - Sanofi-Aventis Administrative Office, Santiago
  - Sanofi-aventis adminsitrative office, Santiago
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, San Juan, Puerto Rico
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden